CLINICAL TRIAL: NCT04705922
Title: A Phase I, Single-Center, Open-Label, 3-Way Crossover, Randomized Single Dose Study to Evaluate the Food Effect on the Pharmacokinetics of TT-00420 Tablet and to Determine the Relative Bioavailability of TT-00420 Tablet Versus TT-00420 Capsule in Adult Healthy Volunteers
Brief Title: Relative Bioavailability Study and Food Effect Study of TT-00420 (Tinengotinib) Capsule and Tablet Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TT420HV1102
Record Dates: First submitted 2021-01-06; First posted 2021-01-12 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sequence 1 [TT-00420 tablet, fed; TT-00420 tablet, fasted; TT-00420 capsule, fasted] (Experimental): Participants will receive a single dose of TT-00420 tablet under fed conditions, followed by a single dose of TT-00420 tablet under fasted conditions, followed by a single dose of TT-00420 capsule under fasted conditions. There will be at least a 14-day wash-out period between each dose.
  Interventions: Drug: TT-00420 Capsule; Drug: TT-00420 Tablet
- Sequence 2 [TT-00420 tablet, fasted; TT-00420 capsule, fed; TT-00420 tablet, fed] (Experimental): Participants will receive a single dose of TT-00420 tablet under fasted conditions, followed by a single dose of TT-00420 capsule under fasted conditions, followed by a single dose of TT-00420 tablet under fed conditions. There will be at least a 14-day wash-out period between each dose.
  Interventions: Drug: TT-00420 Capsule; Drug: TT-00420 Tablet
- Sequence 3 [TT-00420 capsule, fasted; TT-00420 tablet, fed; TT-00420 tablet, fasted] (Experimental): Participants will receive a single dose of TT-00420 capsule under fasted conditions, followed by a single dose of TT-00420 tablet under fed conditions, followed by a single dose of TT-00420 tablet under fasted conditions. There will be at least a 14-day wash-out period between each dose.
  Interventions: Drug: TT-00420 Capsule; Drug: TT-00420 Tablet

INTERVENTIONS:
Drug: TT-00420 Capsule — TT-00420 capsule formulation, administered orally
Drug: TT-00420 Tablet — TT-00420 tablet formulation, administered orally

SUMMARY:
This study is an open-label, 3-way crossover randomized study in adult healthy volunteers to evaluate the relative bioavailability of TT-00420 tablet and capsule formulations and to evaluate food effect on the pharmacokinetics of TT-00420 tablet.

DETAILED DESCRIPTION:
Subjects will be randomized to one of three treatment sequences. Each sequence will contain up to 8 subjects. In each treatment sequence, subjects undergo a baseline/screening period, three treatment periods, and a follow-up visit.

Subjects will be administered a single dose of TT-00420 on Day 1 of either TT-00420 tablet under fed condition, TT-00420 tablet under fasting condition, or capsule under fasting condition and crossed over after at least a 14-day washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 64 years of age inclusive, at the time of signing the informed consent.
2. Body mass index (BMI) between 18 and 32 kg/m2, inclusive, and weighs at least 50 kg.
3. Healthy as determined by the investigator based on medical history, clinical laboratory results (serum chemistry, hematology, urinalysis, and serology), vital sign measurements, 12-lead electrocardiogram (ECG) results, and physical examination findings. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only, if per the investigator discretion, the investigator judges and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
4. Male subjects must not donate sperm starting at Screening, throughout the study period and for at least 90 days after final study drug administration.
5. Male subjects with female sexual partner(s) of reproductive potential may be enrolled if the male:

   1. is documented to be surgically sterile (i.e., successfully vasectomized), or
   2. agrees to use 2 methods of highly effective contraception and agree to refrain from sperm donation from the time of Screening through 90 days post-doseHighly effective includes male condom with spermicide PLUS an effective contraceptive for the female partner that includes: OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring or IUD
6. If female, is of non-childbearing potential, meeting the following requirements:

   1. pre-menopausal with documentation of surgical sterilization (i.e., hysterectomy, bilateral tubal ligation, bilateral oophorectomy, or bilateral salpingectomy at least 3 months prior to study entry), or
   2. post-menopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and with follicle-stimulating hormone (FSH) level ≥ 40 mIU/mL at Screening
7. Able to sign the informed consent and comply with the protocol.

Exclusion Criteria:

1. Any history of clinically serious disease.
2. Any active or unstable clinically significant medical condition as judged by the Investigator.
3. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
4. Hypersensitivity or allergy to any of the study drugs or drugs of similar chemical classes.
5. Hypersensitivity or allergy for components of the prescribed meal
6. Received any investigational drug within 30 days or 5 half-lives(whichever is longer, if known) before the study.
7. Subject who has undergone major surgery ≤ 2 months before study drug administration.
8. Impaired cardiac function including clinically significant arrhythmias or clinically significant abnormality in clinical test, including but not limited to any of the following at Screening and Admission, repeat testing is allowed for verification, at the discretion of the Investigator:

   1. Heart rate < 45 beats per minute (bpm) or > 90 bpm.
   2. Systolic blood pressure (SBP) < 90 mmHg or > 140 mmHg; diastolic blood pressure (DBP) < 50 mmHg or > 90 mmHg.
   3. Average of the 3 QT intervals corrected using Fridericia's formula (QTcF) > 450 milliseconds.
   4. Troponin I at screening > upper limit of normal (ULN).
   5. Second degree or higher Atrioventricular block on ECG.
9. Subject who has a known history of, or a positive test result for, hepatitis B surface antigen (HBsAg), immunoglobulin M (IgM) antibody to hepatitis B core antibody (anti-HBc) (IgM anti-HBc), hepatitis C virus antibody (anti-HCV), or human immunodeficiency virus (HIV) types 1 or 2, or syphilis at Screening.
10. Subject with a history of severe visual diseases; or visual changes including flushing lights, blurry vision, color changes, or other visual changes.
11. Subject who has used prescription or over-the-counter (OTC) medication (other than ≤ 2 g/day paracetamol [acetaminophen] or ≤ 800-mg/day ibuprofen), vitamins, or herbal remedies, within 2 weeks or 5 half-lives (if known) before study drug administration, whichever is longer.
12. Subject who has had a loss of more than 100 mL blood (e.g., a blood donation) within 2 months before study drug administration, or has received any blood, plasma, or platelet transfusions within 3 months before Admission, or plans to donate blood during the study or within 3 months after the study.
13. Subject who has a history of alcohol abuse (defined as an alcohol intake more than 21 units for males and 14 units for females per week) or a history of drug abuse within the 6 months before study drug administration, or a history of substance abuse deemed significant by the Investigator.
14. Subject who smokes cigarettes or uses other nicotine-containing products (e.g., snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers), and has done so in the 3 months prior to Screening.
15. Subject who has a positive test for alcohol or drugs of abuse (opiates, methadone, buprenorphine, methamphetamine, cocaine, cannabinoids, amphetamines, or cotinine) at Screening or Admission.
16. Subject is unable to complete this study for other reasons or the Investigator believes that he or she should be excluded.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-03-07 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC0-∞) of TT-00420 | From pre-dose up to 240 hours post-dose each period (each period is 14 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis of TT-00420.
Area under the curve (AUC0-t) of TT-00420 | From pre-dose up to 240 hours post-dose each period (each period is 14 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis of TT-00420.
Maximum observed concentration (Cmax) of TT-00420 | From pre-dose up to 240 hours post-dose each period (each period is 14 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis of TT-00420.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | From admission up to 10 days following discharge
Incidence of abnormal physical examinations | At baseline and from admission to discharge, up to 12 days per period (each period is 14 days)
Incidence of abnormal clinical laboratory tests | At baseline and from admission to discharge, up to 12 days per period (each period is 14 days)
Incidence of abnormal vital signs | At baseline and from admission to discharge, up to 12 days per period (each period is 14 days)
Incidence of abnormal weight | At baseline and from admission to discharge, up to 12 days per period (each period is 14 days)
Incidence of abnormal 12-lead electrocardiogram | At baseline and from admission to discharge, up to 12 days per period (each period is 14 days)
Half life (t1/2) of TT-00420 | From pre-dose up to 240 hours post-dose each period (each period is 14 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis of TT-00420.
Time of maximum concentration (tmax) of TT-00420 | From pre-dose up to 240 hours post-dose each period (each period is 14 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis of TT-00420.
Volume of distribution (Vd/F) of TT-00420 | From pre-dose up to 240 hours post-dose each period (each period is 14 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis of TT-00420.
Clearance (CL/F) of TT-00420 | From pre-dose up to 240 hours post-dose each period (each period is 14 days)
  Blood samples will be collected at indicated time points for pharmacokinetic analysis of TT-00420.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, Principal Investigator — Pharmaron CPC
Locations (1):
- Pharmaron CPC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No